CLINICAL TRIAL: NCT04128202
Title: Online Intervention to Prevent Perinatal Depression and Promote Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jennifer Duffecy, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0519
Record Dates: First submitted 2019-10-02; First posted 2019-10-16 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Depression; Breastfeeding
MeSH Terms: conditions — Depression; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunnyside (Active Comparator): An online intervention to better manage mood during and after pregnancy.
  Interventions: Behavioral: Sunnyside
- Sunnyside Plus (Experimental): An online intervention to better manage mood and promote and support breastfeeding during and after pregnancy.
  Interventions: Behavioral: Sunnyside Plus

INTERVENTIONS:
Behavioral: Sunnyside — The Sunnyside intervention is an online intervention (an interactive website with didactic material and interactive tools) targeting skills to manage mood during and after pregnancy. The Sunnyside intervention will consist of 6weeks of online lessons during pregnancy and booster sessions at 2 weeks, 4 weeks, and 6 weeks postpartum. Each lesson takes approximately 10 minutes to complete.
  Arms: Sunnyside
Behavioral: Sunnyside Plus — Sunnyside Plus will build upon the Sunnyside intervention, plus include additional education and support to promote breastfeeding. Breastfeeding education and skills will be provided during the 6weeks of online lessons during pregnancy; each lesson takes approximately 10 minutes to complete. Breastfeeding support will continue through 6 weeks postpartum. This postpartum support will involve weekly online lessons(each taking approximately 10 minutes to complete), text support messages(3 sent during weeks 1 and 2, 2 sent during weeks 3 and 4, 1 sent during weeks 5 and 6), and video support calls with a Lactation Educator (LE)provided on an as-needed basis(exception: at least 1 video call is required during both week 1 postpartum and week 2 postpartum).
  Arms: Sunnyside Plus

SUMMARY:
"SunnysidePlus" will functionally integrate a web based intervention targeting skills to promote and support breastfeeding, manage mood,and prevent depression. Sunnyside Plus will build upon the previously tested "Sunnyside" intervention which targeted skills to manage mood through an interactive website with didactic material and tools. Women in weeks 20-28 of their pregnancy will be randomized to receive either Sunnyside Plus or Sunnyside. The Sunnyside intervention will consist of 6 weeks of online lessons during pregnancy and booster sessions at 2 weeks, 4 weeks, and 6 weeks postpartum. Sunnyside Plus will include additional education and support to improve breastfeeding outcomes. Breastfeeding education and skills will be provided during the 6 weeks of online lessons during pregnancy. Breastfeeding support will continue through 6 weeks postpartum. This postpartum support will involve weekly online lessons, text support, and video support calls with a Lactation Educator provided on an as-needed basis. SunnysidePlus has the potential to provide a novel paradigm for improving breastfeeding outcomes and preventing depression; one that is accessible, highly scalable and cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Black or African American
* 18 years and older
* Pregnant and between 20 and 28 weeks gestation
* Intend to breastfeed their child
* Have a score of 5-14 on the Patient Health Questionnaire-8 (PHQ-8)
* Have access to a broadband internet connection
* Are able to read and speak English

Exclusion Criteria:

* Are pregnant with multiples
* Have visual, hearing, voice, or motor impairment that would prevent completion of study procedures
* Diagnosed with a major depressive episode, psychotic disorder, bipolar disorder, dissociative disorder, substance use disorder or other diagnosis for which participation in this trial is either inappropriate or dangerous based on self-report
* Are currently receiving treatment (medication or psychotherapy),have an intention to resume antidepressant medication after delivery (i.e., women who discontinued their medication during pregnancy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 2 weeks
  The PHQ-9 is composed of 9 scored items and 1 unscored item which reflect overall functioning and impairment due to the depressive symptoms. PHQ-9 scoring interpretations are as follows: 1-4: minimal depressive symptoms; 5-9 mild depressive symptoms; 10-14: moderate depressive symptoms; 15-19: moderately severe depressive symptoms: 20-27: severe depressive symptoms.
Breastfeeding Status | Through 12 weeks postpartum
  Breastfeeding initiation, exclusivity, and duration will be assessed in the postpartum period.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Duffecy, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pezley L, Tussing-Humphreys L, Koenig MD, Maki P, Odoms-Young A, Freels S, DiPiazza B, Cann F, Cares K, Depa C, Klejka G, Lima Oliveira M, Prough J, Roe T, Buscemi J, Duffecy J. Feasibility of a Web-Based Intervention to Prevent Perinatal Depression and Promote Human Milk Feeding: Randomized Pilot Trial. JMIR Form Res. 2022 May 3;6(5):e32226. doi: 10.2196/32226. PMID 35503244